CLINICAL TRIAL: NCT02386514
Title: Emergency Department, Rapid Assessment for Sexually Transmitted Infection
Acronym: ED-RASTI
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Principal Investigator, Joseph Miller, MD, Clinical Physician, Henry Ford Health System
Other Study IDs: 9107
Record Dates: First submitted 2015-01-09; First posted 2015-03-12 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Infection
Keywords: sexually transmitted infection; gonorrhea; chlamydia; presumptive therapy
MeSH Terms: conditions — Infections; Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate if a rapid urine Nucleic Acid Amplification Testing (NAAT) is non-inferior to the traditional swab NAAT for gonorrhea and chlamydia when performed in the Emergency Department.

DETAILED DESCRIPTION:
All patients presenting to the Emergency Department during the study period who are tested for gonorrhea and chlamydia by the traditional swab NAAT will concurrently have their urine tested for gonorrhea and chlamydia using the Cepheid GeneXpert rapid NAAT. The result of both tests will be compared to determine if the rapid assay is non-inferior to the current traditional NAAT. Both the traditional and Cepheid GeneXpert rapid NAAT are FDA and CDC approved for evaluation of gonorrhea and chlamydia. However, the Cepheid GeneXpert rapid NAAT has not been prospectively validated in the Emergency Department setting. We intend for both the provider obtaining the sample and the technician running the rapid assay sample to be blinded to the result of the traditional NAAT. The Cepheid GeneXpert rapid NAAT will not be used in patient care decisions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical concern for gonorrhea and/or chlamydia infection
* Concurrent testing for gonorrhea and chlamydia using traditional NAAT assay

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients greater than 18 years of age presenting with a complaint that triggers the providing clinician to obtain a gonorrhea and chlamydia test by the traditional format.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of a chlamydia trachomatis or neisseria gonorrhoeae | 24 hours
  comparative test characteristics to traditional swab in the Emergency Department.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Derived] Wilson SP, Vohra T, Goldberg J, Price C, Calo S, Mahan M, Miller J. Reliable Rapid Assay for Gonorrhea and Chlamydia in the Emergency Department. J Emerg Med. 2017 Dec;53(6):890-895. doi: 10.1016/j.jemermed.2017.08.094. Epub 2017 Oct 23. PMID 29074030